CLINICAL TRIAL: NCT06129747
Title: Repeat Breast Conserving Surgery Followed by Daily Partial Breast Irradiation for Participants With Ipsilateral Breast Tumor Recurrence Treated Initially With Breast Conserving Surgery and Whole Breast Radiation Therapy
Brief Title: Repeat Breast Conserving Surgery Followed by Daily Partial Breast Irradiation in Ipsilateral Breast
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4123
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Tumor, Breast
Keywords: Radiation Therapy; In-Breast Recurrence; Tumor; Re-irradiation
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Participants will receive once daily radiation for 15 fractions to 40.05 Gy total dose. Participants with high risk features (high grade disease, young age, close margins (<2mm), triple negative subtype, HER2 positive tumors not receiving HER2 targeted systemic therapy) may receive a simultaneous boost to 48 Gy in 15 fractions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy(RT) (Experimental): There will be one treatment cohort. Radiation therapy will be delivered daily for 15 daily fractions, 2.67Gy per fraction, delivered using a 3-D or IMRT(Intensity Modulate Radiation Therapy) plan. For participants with high-risk features deemed by the radiation oncologist who would otherwise be a candidate for a boost (age <50, high grade, poor biology, close margins), 48 Gy delivered in fifteen fractions of 3.2 Gy is allowed.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Weeks 1, 2 and 3
  * Weeks 1, 2 and 3 will include 5 days of treatment.
  * One radiation treatment to breast on each of the 5 days. Each radiation treatment session will last a 30 minutes.

SUMMARY:
The standard treatment for participants whose cancer has returned after breast conserving surgery is radiation given twice daily (separated by at least 6 hours) for a total of 30 treatments. The purpose of this study is to find out if giving radiation once a day for 15 treatments after repeat breast conserving surgery works as well as giving it the standard way.

DETAILED DESCRIPTION:
Breast cancer survival rates have greatly improved with advances in both screening and treatment. The standard of care for both early stage and selected locally advanced breast cancers is breast conserving therapy (BCT), consisting of a partial mastectomy followed by radiation treatment. Traditionally, a salvage mastectomy was the standard treatment for women who initially underwent BCT and experienced an ipsilateral breast tumor recurrence (IBTR). Many participants have become increasingly motivated to avoid mastectomy, and there has been rising interest in repeat BCS (Breast Conserving Surgery) with focal radiation for certain participants motivated to keep their breast. The current standard of care for breast re-irradiation after an in-breast tumor recurrence is partial breast irradiation consisting of a dose of 45 Gy delivered BID for 30 fractions. While this regimen demonstrated excellent local control and low AEs, the regimen itself is difficult for participants. Receiving RT twice daily at smaller doses per fraction (1.5 Gy) for 30 treatments can be burdensome, especially for those without reliable transportation or difficulty getting time away from work. Given the excellent local control rates and low rate of AEs, in this study, we hypothesize that daily hypofractionated EBRT(External Beam Radiation Therapy) for re-irradiation after repeat BCS would be at least as well tolerated with good local control and provide a more convenient option for participants than the current standard of care established by RTOG 1014. Some participants will present with high-risk features (e.g. age <50, high grade, ER negative tumors, close margins) making dose escalation an attractive option to improve local control. Options for dose escalation include sequential and concurrent administration of a boost.

ELIGIBILITY:
Inclusion Criteria:

* Participants' recurrences must have histologically confirmed ductal carcinoma in-situ, invasive ductal, medullary, papillary, colloid (mucinous), tubular or mixed histologies. Three years of time must have elapsed since the end of the last course of whole breast irradiation.
* Lesion size < 3 cm treated with a partial mastectomy. Participants with invasive cancer and clinically and radiographically negative axillas do not require an axillary lymph node sampling unless they did not have prior axillary lymph node sampling (e.g. previous cancer was DCIS). Participants with DCIS as their recurrence do not require surgical assessment of the axilla. Repeat sentinel lymph node biopsy is permitted.
* Negative resection margins with at least no tumor on ink or a negative re-excision.
* Participants with invasive recurrence must have a negative re-staging work-up consisting of either a CT chest/abdomen and a bone scan or a PET scan.
* Hormonal therapy is allowed. If chemotherapy is planned, it can be delivered either prior to or after the radiation is delivered. There must be at least 2 weeks between radiation and chemotherapy. HER2 directed therapy can be delivered concurrently with radiation.
* Participants must be > 18 years of age. Because no dosing or adverse event data are currently available on the use of breast re-irradiation in participants ≤18 years of age, children are excluded from this study.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Performance status: ECOG Performance status ≤ 2.
* Life expectancy of ≥ 12months, in the opinion of and as documented by the investigator.
* Not based on gender; this trial is open to any gender, defined as self-representation of gender identity.

Exclusion Criteria:

* Participants with nodal or distant metastatic disease < 3 years since prior radiation.
* Participants with invasive pure lobular carcinoma, extensive lobular carcinoma in-situ, extensive ductal carcinoma in-situ (spanning more than 3 cm), or uncontrolled nonepithelial breast malignancies such as lymphoma or sarcoma.
* Participants with multicentric carcinoma (tumors in different quadrants of the breast or tumors separated by at least 4 cm). Palpable or radiographically suspicious contralateral axillary, ipsilateral or contralateral supraclavicular, infraclavicular, or internal mammary lymph nodes unless these are histologically or cytologically confirmed negative.
* Participants with Paget's disease of the nipple.
* Participants with skin involvement.
* Participants with scleroderma or dermatomyositis.
* Participants with psychiatric, neurologic, or addictive disorders that would preclude obtaining informed consent.
* Participants who are pregnant or lactating due to potential fetal exposure to radiation and unknown effects of radiation on lactating females.
* Participants with known BRCA 1/BRCA 2 mutations.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2029-08-09 (Estimated); Study Completion 2029-08-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events as graded by CTCAE criteria | 1 year from the completion of re-irradiation
  Rate of grade 3+ treatment-related skin, fibrosis, and breast pain adverse events occurring within 1 year from the completion of re-irradiation as graded by CTCAE criteria.

SECONDARY OUTCOMES:
In-breast tumor recurrence rate | 3 years
  The overall in-breast tumor recurrence rate will be estimated using the cumulative incidence function.
In-breast tumor recurrence rate | 5 years
  The overall in-breast tumor recurrence rate is estimated using the cumulative incidence function.
In-breast tumor recurrence rate | 10 years
  The overall in-breast tumor recurrence rate will be estimated using the cumulative incidence function.
Rate of freedom from mastectomy | 3 years
  The freedom from mastectomy rate will be estimated using the cumulative incidence function.
Rate of freedom from mastectomy | 5 years
  The freedom from mastectomy rate will be estimated using the cumulative incidence function.
Rate of freedom from mastectomy | 10 years
  The freedom from mastectomy rate will be estimated using the cumulative incidence function.
Treatment-related adverse events | 1 year from completion of re-irradiation
  All treatment-related adverse events for the defined time periods
Treatment-related adverse events | Overall for 3 years from completion of re-irradiation
  All treatment-related adverse events for the defined time periods
Evaluation of Cosmesis | 1 year
  Determined by an established Global Cosmesis Score grading from 1 through 4, with 1 being excellent and 4 being rated as poor
Evaluation of Cosmesis | 3 years
  Determined by an established Global Cosmesis Score grading from 1 through 4, with 1 being excellent and 4 being rated as poor
Overall survival rate | 3 years
  Overall survival will be estimated using Kaplan-Meier Method
Overall survival rate | 5 years
  Overall survival will be estimated using Kaplan-Meier Method
Overall survival rate | 10 years
  Overall survival will be estimated using Kaplan-Meier Method
Mastectomy-free survival rate | 3 years
  Mastectomy-free survival will be estimated using Kaplan-Meier Method
Mastectomy-free survival rate | 5 years
  Mastectomy-free survival will be estimated using Kaplan-Meier Method
Mastectomy-free survival rate | 10 years
  Mastectomy-free survival will be estimated using Kaplan-Meier Method

CONTACTS AND LOCATIONS:
Overall Officials: Janice Lyons, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Rahul Tendulkar, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Data will be used for study purposes only and not otherwise shared